CLINICAL TRIAL: NCT05665413
Title: Effects of Stroking Versus Ergon Technique on Lateral Cutaneous Femoral Nerve Radiculopathy and Functional Activity in Pregnant Women
Brief Title: Stroking Versus Ergon Technique in Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/22/0542 Sadaf Anjum
Record Dates: First submitted 2022-12-17; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Lateral Cutaneous Nerve of Thigh Lesion
Keywords: numbness; thigh; pain
MeSH Terms: conditions — Hypesthesia; Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- strocking technique (Experimental)
  Interventions: Device: TENS
- ergon technique (Experimental)
  Interventions: Device: TENS

INTERVENTIONS:
Device: TENS — strocking technique, HOT PACK and Ergon instrument
  Other Names: HOT PACK; Ergon instrument; strocking technique

SUMMARY:
The study will focus on non-invasive management options for radiculopathy and functional activity in 3rd trimester women due to lateral cutaneous femoral nerve study. The findings of this study will help future clinicians to develop management plans for these patients that can include non-invasive and non-pharmacological treatment options like Ergon Technique and Stroking based on their effectiveness. The lateral femoral cutaneous nerve is formed by posterior divisions of the anterior rami of spinal nerves to enter the iliac fossa. It continues into the anterolateral thigh by passing either below or through the inguinal ligament, emerging anterior to the Sartorius muscle L2 and L3 In the thigh, it gives rise to two branches, The anterior branch supplies the skin of the anterolateral thigh to the knee and the posterior branch innervates the skin of the lateral aspect of the greater trochanter to the mid-thigh region. It can be compressed due to swelling, trauma or pressure in the surrounding areas. Common causes may include: Tight clothing, obesity or weight gain, and pregnancy. Symptoms may include anterior and lateral thigh burning, tingling, and numbness.

It will be a randomized clinical trial aimed to find the comparative effects of stroking and ergon technique on radiculopathy and functional activity in pregnant women. Women who meet the inclusion criteria that is they show positive femoral traction test, two point discrimination, light touch and pin prick maneuver will be recruited from Surya Azeem Hospital and Jinnah Hospital, Lahore. Two groups will be formed 13 patients will be allocated in each group. Before applying the techniques pre treatment reading will taken after that Hot Pack and TENS will be applied as a baseline treatment to both groups while Ergon technique will be applied to group A while stroking will be applied to the patients of group B. Two sessions per week will be given for 8 weeks. After that post treatment reading will be taken on 8th week. Data will be analyzed by using SPSS for windows version 25

ELIGIBILITY:
Inclusion Criteria:

* Pregnant ladies during 3rd trimester.
* Pregnant ladies of age between 30 to 40 years.
* Primigravida and Multigravida ladies.

Exclusion Criteria:

* Pregnant ladies with any previous hip fracture.
* Women with high risk pregnancy.
* Any previous history of disc herniation.
* Patients with lumbar radiculopathy.

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only pregnant women
Enrollment: 24 (Estimated)
Dates: Start 2021-12-24 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Pain DETECT questionnaire PDQ | 8th week
  painDETECT (PDQ) is a symptom-based assessment tool. It is a nine-item questionnaire that consists of seven sensory symptom items for pain that are graded from 0= never to 5= strongly, one temporal item on pain-course pattern graded -1 to +1, and one spatial item on pain radiation graded 0 for no radiation or +2 for radiating pain. Total scoring is 35.
The Lower Extremity Functional Scale (LEFS) | 8th week
  The Lower Extremity Functional Scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used by clinicians as a measure of patients' initial function, ongoing progress and outcome, as well as to set functional goals.Total scoring is 80.

CONTACTS AND LOCATIONS:
Overall Officials: fatima tariq, TDPT, Study Chair — Riphah International University
Locations (1):
- Surya Azeem Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No